CLINICAL TRIAL: NCT06131957
Title: Root Caries Prevention Using Fluoride Varnish Fortified With Strontium-doped Bioactive Glass Ceramic: a Randomized Double-blind Controlled Clinical Trial
Brief Title: Root Caries Prevention Using Fluoride Varnish Fortified With SBGC
Acronym: SBGC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UW23-451
Record Dates: First submitted 2023-11-08; First posted 2023-11-15 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-01

CONDITIONS: Dental Caries of Root Surface; Root Caries
Keywords: Strontium-doped Bioactive Glass Ceramic; Fluoride varnish; Older adults; Root caries; Dentine; Prevention
MeSH Terms: conditions — Root Caries | interventions — sodium fluoride topical preparation

STUDY DESIGN:
Intervention Model Description: Participants are randomized assigned to either experimental group or controlled group.
Who Masked: Participant, Investigator
Masking Description: The subjects and the clinical team including the dentist and the dental surgery assistant will all be blinded to the subjects' assignment of the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoride varnish with SBGC (Experimental): This group will receive applications of fluoride varnish (containing 5% NaF) with 7.5% SBGC every 3 months for 36 months.
  Interventions: Combination Product: Fluoride varnish with SBGC
- Fluoride varnish without SBGC (Active Comparator): This group will receive 5% NaF varnish with SBGC every 3 months for 36 months.
  Interventions: Drug: Fluoride varnish

INTERVENTIONS:
Combination Product: Fluoride varnish with SBGC — The Fluoride varnish (containing 5% NaF, Duraphat®, Colgate-Palmolive Company, NY, USA) mixed with 7.5% SBGC (Dencare (Chongqing) Oral Care Co., Ltd).
  Arms: Fluoride varnish with SBGC
Drug: Fluoride varnish — The Fluoride varnish (containing 5% NaF, Duraphat®, Colgate-Palmolive Company, NY, USA)
  Other Names: Duraphat
  Arms: Fluoride varnish without SBGC

SUMMARY:
The goal of this 36-month double-blind randomized controlled trial is to compare the effects of 5% sodium fluoride varnish (22,600 ppm fluoride) with or without Strontium-doped bioactive glass (SBGC) on root caries development in community-dwelling older adults.

DETAILED DESCRIPTION:
This 36-month, double-blind, two-arm randomized controlled trial is aimed to compare the effects of 5% sodium fluoride varnish (22,600 ppm fluoride) with or without Strontium-doped bioactive glass (SBGC) on root caries development in community-dwelling older adults.

Participants will be divided in to two groups, The main question it aims to answer is: Is fluoride varnish with SBGC more effective than that without SBGC on prevention root caries in community-dwelling older adults? Participants will be divided into two groups, experimental group and controlled group after randomization. Subjects in the experimental group will receive fluoride varnish with SBGC quarterly, and subjects in the controlled group will receive fluoride varnish without SBGC quarterly.

It is hypothesized that community-dwelling older adults who receive quarterly fluoride varnish applications containing SBGC will develop fewer root caries.

ELIGIBILITY:
Inclusion Criteria:

* Adult > 60 years old
* good collaborative relationships

Exclusion Criteria:

* less than 8 natural teeth
* have severe medical conditions
* are in use of high fluoride toothpaste

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
New root caries lesions and restorations | Baseline, 12, 24, 36 months
  All exposed root surfaces will be examined for new caries lesions based on the ICDAS criteria. Restorations due to root caries will also be recorded after confirmation with the subjects.

SECONDARY OUTCOMES:
Arrested root caries | Baseline, 12, 24, 36 months
  An active root caries lesion found at baseline changed into inactive at follow-ups, according to ICDAS II criteria.
Satisfaction of the use of varnish | 12, 24, 36 months
  Investigated by survey.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine CM Leung, BDS,MDS,PhD, Principal Investigator — Faculty of Dentistry, The University of Hong Kong
Locations (1):
- Clinical Research Center, the Prince Philips Dental Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No